CLINICAL TRIAL: NCT00284908
Title: Pharmacodynamic Dose-Response of S-Tenatoprazole-Na (STU-Na) 30 mg, 60 mg, 90 mg and 120 mg in Healthy Volunteers
Brief Title: Dose-Effect of S-Tenatoprazole-Na(STU-Na) 30 mg, 60 mg, 90 mg and 120 mg in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: STEBA France (Industry)
Collaborators: STEBA LABORATORIES LTD. (Unknown)
Responsible Party: Christof Kreutz/Project leader, STEBA France
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HPD/STU(-Na) 05819N/TU 1.41
Record Dates: First submitted 2006-01-31; First posted 2006-02-01 (Estimated); Last update posted 2008-03-24 (Estimated); Status verified 2008-03

CONDITIONS: Esophagitis; Gastroesophageal Reflux; Stomach Ulcer; Duodenal Ulcer
Keywords: S-Tenatoprazole-Na; Pharmacokinetic; intragastric pH recording; dose-response
MeSH Terms: conditions — Esophagitis; Gastroesophageal Reflux; Stomach Ulcer; Duodenal Ulcer

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- I STU-Na (Experimental): Cross-over study with escalating doses
  Interventions: Drug: S-Tenatoprazole-Na (STU-Na)

INTERVENTIONS:
Drug: S-Tenatoprazole-Na (STU-Na) — 30 mg, 60 mg, 90 mg and 120 mg of STU-Na for 5 days every morning

SUMMARY:
S-Tenatoprazole-Na (STU-Na), a new drug currently under clinical development, belongs to a class of drugs, called proton pump inhibitors (PPls). Some PPIs are already commercially available. STU-Na will be used for treatment of acid related diseases (gastroduodenal ulcers, erosive or ulcerative esophagitis due to gastroesophageal reflux disease). This study evaluates the degree of acid suppression by different doses of STU-Na. The degree of acid suppression is considered to be correlated with clinical efficacy.

In this study four dosages of STU-Na (30 mg, 60 mg, 90 mg, and 120 mg) will be tested in each volunteer. First, one of the dosages will be orally administered for five days. Then, a nine to sixteen day period without study drug administration will follow prior to the administration of the next dosage, for again five days. Each volunteer will have a total of four study drug administration periods.

After the last study drug intake in period 1, 2 and 3 pharmacokinetic blood sampling will be done for four days. After the last study drug intake in period 4 pharmacokinetic blood sampling will be done for five days. Pharmacokinetic blood sampling consists of several blood draws over a pre-determined time period. The pharmacokinetic blood sampling measures the medication concentration in the blood at pre-defined time points.

After the last study drug intake in period 1, 2, 3, and 4, gastric acidity will be measured for 24 hours by means of a thin tube that will be inserted into the stomach through the nostril to evaluate the efficacy of the different dosages of STU-Na.

DETAILED DESCRIPTION:
S-Tenatoprazole-Na (STU-Na), a new drug currently under clinical development, belongs to a class of drugs, called proton pump inhibitors (PPls). Some PPIs are already commercially available. STU-Na will be used for treatment of acid related diseases (gastroduodenal ulcers, erosive or ulcerative esophagitis due to gastroesophageal reflux disease). This study evaluates the degree of acid suppression by different doses of STU-Na. The degree of acid suppression is considered to be correlated with clinical efficacy.

In this study four dosages of STU-Na (30 mg, 60 mg, 90 mg, and 120 mg) will be tested in each volunteer. First, one of the dosages will be orally administered for five days. Then, a nine to sixteen day period without study drug administration will follow prior to the administration of the next dosage, for again five days. Each volunteer will have a total of four study drug administration periods.

After the last study drug intake in period 1, 2 and 3 pharmacokinetic blood sampling will be done for four days. After the last study drug intake in period 4 pharmacokinetic blood sampling will be done for five days. Pharmacokinetic blood sampling consists of several blood draws over a pre-determined time period. The pharmacokinetic blood sampling measures the medication concentration in the blood at pre-defined time points.

After the last study drug intake in period 1, 2, 3, and 4, gastric acidity will be measured for 24 hours by means of a thin tube that will be inserted into the stomach through the nostril to evaluate the efficacy of the different dosages of STU-Na.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers aged 18 to 55 years inclusive
* Able to understand the nature of the study and to give written informed consent
* Able to communicate well with the investigator himself or his/her representatives
* Able not to smoke during each hospitalization
* Normal physical examination at the screening visit
* Body Mass Index between 18 kg/m² and 35 kg/m² at the screening visit
* Normal blood pressure and heart rate measured under standardized conditions at the screening visit after at least 5 minutes of rest in a supine position: SBP within 90 and 140 mmHg, DBP within 40 and 85 mmHg, and HR within 40 to 85 bpm
* Normal 12-lead electrocardiogram at screening visit recorded after at least 5 minutes of rest: PR within 120 and 200 ms, QRS below or equal to 120 ms, and QTc below or equal to 440 ms
* Laboratory results within the normal ranges or considered not being of clinical relevance by the investigator

Exclusion Criteria:

* Vegetarians
* Positive to H. pylori by 13C urea breath test or stool antigen test at screening visit
* Contra-indication to proton pump inhibitors treatment
* Previous participation in a trial with PPIs within 3 months
* Current or historical evidence of clinically relevant cardiovascular, neurological, hematological, hepatic, gastrointestinal, renal, pulmonary, endocrinological, metabolic or psychiatric disease
* Any other acute or chronic disease which could influence the volunteer's health and/or the study results
* Presence or history of malabsorption or any gastrointestinal surgery except appendectomy or hernia repair
* Receipt of medication (including 'over the counter' preparations) within two weeks of dosing
* Use of enzyme inducers or enzyme inhibitor drugs within the last three months before the first drug administration
* Participation in a clinical trial involving receipt of a licensed (marketed) medicinal product or of an unlicensed (investigational) medicinal product within one month before the study
* Past or current drug exposure amounting to drug abuse or addiction
* Past or current alcohol exposure amounting to alcohol abuse or addiction; (i.e. > 28 units per week for males, where 1 unit = one measure of spirit (25 mL), one glass of wine (125 mL) or ½ pint beer)
* Currently smoke >10 cigarettes per day
* Donation of blood or any other major blood loss (>500 mL) within three months before the study
* Unwilling or unable to comply with the study protocol for any reason or in the opinion of the investigator should not participate in the study
* Positive test for hepatitis B surface antigen, hepatitis C antibody, HIV1 or HIV2 antibody at screening
* Known allergy or intolerance to lactose
* Known allergy or intolerance to any other compound in the study drug or any other closely related compound

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2006-09; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Intragastric pH recording for 24 hours after 5 days of treatment | Beginning of the pH recording before the last study drug intake in each period

SECONDARY OUTCOMES:
Pharmacokinetic blood sampling at steady state | Blood sampling begins before the intake of the last study drug in each period and lasts for 96 hours (periods 1 to 3) or 120 hours (period 4)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis A Ruff, MD, Principal Investigator — Healthcare Discoveries Inc.; Patrick Cohen, MD, Study Director — STEBA France; Christof Kreutz, MD, Study Director — STEBA France
Locations (1):
- Healthcare Discoveries, Inc., San Antonio, Texas, United States

REFERENCES:
- [Background] Burget DW, Chiverton SG, Hunt RH. Is there an optimal degree of acid suppression for healing of duodenal ulcers? A model of the relationship between ulcer healing and acid suppression. Gastroenterology. 1990 Aug;99(2):345-51. doi: 10.1016/0016-5085(90)91015-x. PMID 2142113
- [Background] DeVault KR, Castell DO. Updated guidelines for the diagnosis and treatment of gastroesophageal reflux disease. The Practice Parameters Committee of the American College of Gastroenterology. Am J Gastroenterol. 1999 Jun;94(6):1434-42. doi: 10.1111/j.1572-0241.1999.1123_a.x. No abstract available. PMID 10364004
- [Background] Armstrong D. Review article: gastric pH -- the most relevant predictor of benefit in reflux disease? Aliment Pharmacol Ther. 2004 Oct;20 Suppl 5:19-26; discussion 38-9. doi: 10.1111/j.1365-2036.2004.02140.x. PMID 15456460
- [Background] Bell NJ, Burget D, Howden CW, Wilkinson J, Hunt RH. Appropriate acid suppression for the management of gastro-oesophageal reflux disease. Digestion. 1992;51 Suppl 1:59-67. doi: 10.1159/000200917. PMID 1397746
- [Background] Galmiche JP, Bruley Des Varannes S, Ducrotte P, Sacher-Huvelin S, Vavasseur F, Taccoen A, Fiorentini P, Homerin M. Tenatoprazole, a novel proton pump inhibitor with a prolonged plasma half-life: effects on intragastric pH and comparison with esomeprazole in healthy volunteers. Aliment Pharmacol Ther. 2004 Mar 15;19(6):655-62. doi: 10.1111/j.1365-2036.2004.01893.x. PMID 15023167
- [Background] Horn J. The proton-pump inhibitors: similarities and differences. Clin Ther. 2000 Mar;22(3):266-80; discussion 265. doi: 10.1016/S0149-2918(00)80032-6. PMID 10963283
- [Background] Kakinoki B, Ono C, Yamazaki N, Chikamatsu N, Wakatsuki D, Uchiyama K, Morinaka Y. General pharmacological properties of the new proton pump inhibitor (+/-)-5-methoxy-2-[[(4-methoxy-3,5-dimethylpyrid-2-yl)methyl]sulf inyl]- 1H-imidazo[4,5-b]pyridine. Methods Find Exp Clin Pharmacol. 1999 Apr;21(3):179-87. doi: 10.1358/mf.1999.21.3.534827. PMID 10389120
- [Background] Katz PO, Castell DO, Chen Y, Andersson T, Sostek MB. Intragastric acid suppression and pharmacokinetics of twice-daily esomeprazole: a randomized, three-way crossover study. Aliment Pharmacol Ther. 2004 Aug 15;20(4):399-406. doi: 10.1111/j.1365-2036.2004.02079.x. PMID 15298633
- [Background] Kromer W, Horbach S, Luhmann R. Relative efficacies of gastric proton pump inhibitors: their clinical and pharmacological basis. Pharmacology. 1999 Aug;59(2):57-77. doi: 10.1159/000028306. PMID 10450061
- [Background] Lundell LR, Dent J, Bennett JR, Blum AL, Armstrong D, Galmiche JP, Johnson F, Hongo M, Richter JE, Spechler SJ, Tytgat GN, Wallin L. Endoscopic assessment of oesophagitis: clinical and functional correlates and further validation of the Los Angeles classification. Gut. 1999 Aug;45(2):172-80. doi: 10.1136/gut.45.2.172. PMID 10403727
- [Background] Revicki DA, Crawley JA, Zodet MW, Levine DS, Joelsson BO. Complete resolution of heartburn symptoms and health-related quality of life in patients with gastro-oesophageal reflux disease. Aliment Pharmacol Ther. 1999 Dec;13(12):1621-30. doi: 10.1046/j.1365-2036.1999.00669.x. PMID 10594397
- [Background] Stedman CA, Barclay ML. Review article: comparison of the pharmacokinetics, acid suppression and efficacy of proton pump inhibitors. Aliment Pharmacol Ther. 2000 Aug;14(8):963-78. doi: 10.1046/j.1365-2036.2000.00788.x. PMID 10930890
- [Background] Uchiyama K, Wakatsuki D, Kakinoki B, Takeuchi Y, Araki T, Morinaka Y. The long-lasting effect of TU-199, a novel H+, K(+)-ATPase inhibitor, on gastric acid secretion in dogs. J Pharm Pharmacol. 1999 Apr;51(4):457-64. doi: 10.1211/0022357991772510. PMID 10385219